CLINICAL TRIAL: NCT01407731
Title: Analysis of Intersectin Expression in Primary Human Neuroblastomas
Brief Title: Protein Expression in Human Neuroblastoma Tumor Samples
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL11B4; COG-ANBL11B4 (Other: Children's Oncology Group); ANBL11B4 (Other: Children's Oncology Group); NCI-2011-03799 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-07-30; First posted 2011-08-02 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; localized resectable neuroblastoma; localized unresectable neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Blotting, Western

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: protein expression analysis
Genetic: western blotting
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying protein expression in samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat neuroblastoma.

PURPOSE: This laboratory studying is looking at protein expression in tumor tissue samples from patients with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether intersectin (ITSN1) proteins are present at elevated levels in primary human tumor samples.

OUTLINE: Archived tumor tissue samples are analyzed for intersectin (ITSN1) expression by western blot assays with enhanced chemiluminescence and exposed to X-ray film. The films are scanned, and levels of ITSN1 signal are quantified by densitometry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with neuroblastoma
* Banked primary tumor samples from patients with stage 1, 2, 3, and 4 disease

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosed with neuroblastoma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
ITSN1 is highly expressed in neuroblastoma tumors and plays an important role in the development/progression of these tumors

CONTACTS AND LOCATIONS:
Overall Officials: John P. O'Bryan, PhD, Principal Investigator — University of Illinois at Chicago